CLINICAL TRIAL: NCT06065098
Title: Church-based Health Intervention to Eliminate Racial Inequalities in Cardiovascular Health
Acronym: CHERISH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-703-SPHTM
Record Dates: First submitted 2023-08-21; First posted 2023-10-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases; Hypertension; Diabetes; Hypercholesterolemia
Keywords: health inequities; cardiovascular health; community-based interventions; cardiovascular disease prevention
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Diabetes Mellitus; Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: Cluster-randomization of 46 churches in New Orleans, Louisiana to two arms
Who Masked: Outcomes Assessor
Masking Description: Clinical research coordinators and laboratory technicians who assess health-related outcomes will be blinded to intervention assignment. Study physicians who review serious adverse events and unanticipated problems will also be blinded to intervention assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community health worker-led implementation strategy: (Experimental): Individual coaching sessions; healthcare navigation; healthcare at community settings; church-based nutrition education and exercise programs; and self-monitoring of BP.
  Interventions: Behavioral: Evidence-based interventions recommended by the 2019 ACC/AHA Guideline on the Primary Prevention of CVD
- Group-based Education Strategy (Experimental): Group-based education sessions; information on primary care physicians; and instruction on self-monitoring of BP.
  Interventions: Behavioral: Evidence-based interventions recommended by the 2019 ACC/AHA Guideline on the Primary Prevention of CVD

INTERVENTIONS:
Behavioral: Evidence-based interventions recommended by the 2019 ACC/AHA Guideline on the Primary Prevention of CVD — The recommended evidence-based interventions include therapeutic lifestyle change and medical treatment of hypertension, diabetes, and hypercholesterolemia.

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death in the US general population. Although CVD mortality rates declined for both Black and White populations during the past two decades, they are still higher in Black adults than White adults. There are also persistent disparities in CVD risk factors with higher prevalence of obesity, hypertension, and diabetes in Black compared to White populations. In addition, CVD and risk factors are more prevalent in the residents of Louisiana compared to the US general population. The Church-based Health Intervention to Eliminate Racial Inequalities in Cardiovascular Health (CHERISH) study will use a church-based community health worker (CHW)-led multifaceted intervention to address racial inequities in CVD risk factors in predominantly Black communities in New Orleans, Louisiana. The primary aim of the CHERISH study is to compare the impact of two implementation strategies - a CHW-led multifaceted strategy and a group-based education strategy - for delivering interventions recommended by the 2019 American College of Cardiology (ACC)/American Heart Association (AHA) Guideline on the Primary Prevention of Cardiovascular Disease on implementation and clinical effectiveness outcomes in predominantly Black church community members over 18 months.

DETAILED DESCRIPTION:
Louisiana residents, especially African Americans, bear a disproportionately high burden of CVD. In the CHERISH cluster randomized trial, we will compare the impact of two implementation strategies - a CHW-led multifaceted strategy and a group-based education strategy - for delivering interventions recommended by the 2019 ACC/AHA Guideline on the Primary Prevention of Cardiovascular Disease on implementation and clinical effectiveness outcomes in Black community members over 18 months. The CHERISH study utilizes an effectiveness-implementation hybrid design to: (1). test the effectiveness of a CHW-led church-based multifaceted implementation strategy for reducing estimated CVD risk over 18 months among African Americans at high risk for CVD, and (2). assess the implementation outcomes (acceptability, adaptation, adoption, feasibility, fidelity, penetrance, cost-effectiveness, and sustainability) simultaneously. The Exploration, Preparation, Implementation, Sustainment (EPIS) framework has guided the development and evaluation of the multifaceted implementation strategy, which includes CHW-led health coaching on lifestyle changes and medication adherence; healthcare delivery in community; church-based exercise and weight loss programs; self-monitoring of blood pressure (BP); and provider education and engagement. The CHW-led church-based intervention will provide strong social support and tackle multiple social determinants of CVD disparities. The primary effectiveness outcome is change in the estimated 10-year risk for atherosclerotic CVD (ASCVD) using the ACC/AHA Pooled Cohort Equations. The primary implementation outcome is a fidelity summary score for key implementation strategy components during the 18-month intervention. Our study has 96% statistical power to detect a slope difference of 0.83% in 10-year ASCVD risk over 18 months using a 2-sided significance level of 0.05. We will recruit 806 participants (17.5 per church) aged ≥40 years who have <3 ideal cardiovascular health matrices and randomly assign 23 churches to intervention and 23 to control; we will implement the multifaceted intervention program; we will follow-up participants and collect data on effectiveness and implementation outcomes at 6, 12, and 18 months; we will evaluate the sustainability of the intervention at 6 months post-intervention; and we will perform intention-to-treat analyses and disseminate and scale-up the proven-effective implementation strategy. The proposed study will generate evidence on the effectiveness, implementation, and sustainability of the multifaceted intervention aimed at eliminating CVD disparities in predominantly African American communities in the US.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged ≥40 years
* Community members associated with the participating churches (church members and their families and friends)
* Individuals with three or more CVD risk factors (out of seven):

  * Current smoker
  * Overweight or obese (BMI ≥25 kg/m2)
  * Insufficient physical activity (<150 minutes/week moderate intensity or <75 minutes/week vigorous intensity)
  * Healthy diet score of <4 components
  * Total cholesterol ≥200 mg/dL
  * Blood pressure ≥130/80 mmHg
  * Fasting plasma glucose ≥100 mg/dL
* Willing and able to participate in the intervention

Exclusion Criteria:

* No prior hospitalization in the last 3 months for chronic heart failure or heart attack.
* No current diagnosis of cancer requiring chemotherapy or radiation therapy
* No stage-5 chronic kidney disease requiring chronic dialysis, or transplant.
* Not pregnant or planning to become pregnant in the next 18 months.
* No plans to move out of the New Orleans metropolitan area during the next year.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 806 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Difference in change in estimated atherosclerotic cardiovascular disease (ASCVD) risk score | Measured from baseline to 18 months
  The ACC/AHA ASCVD risk score will be calculated using the pooled population cohort equation based on age (years), total cholesterol (mg/dL), high-density lipoprotein (HDL)-cholesterol (mg/dL), antihypertensive medication use, systolic BP (mmHg), current smoking status, and diabetes status. The risk score ranges from 0% to 100%.
Fidelity summary score | Measured at 6, 12, and 18 months
  The fidelity summary score is composed of the following key implementation strategy components: proportion of assigned health education sessions attended in all participants, proportion of assigned discussion sessions attended in all participants, proportion of recommended minutes of physical activity completed in all participants, proportion of days per week that fruits/vegetables are eaten as recommended in all participants, proportion of recommended home BP monitoring completed in patients with hypertension, proportion of required provider visits attended in all patients, and proportion of antihypertensive, antidiabetic, and statin medications taken in patients with hypertension or diabetes, or those who are eligible for statin treatment, respectively.

SECONDARY OUTCOMES:
Difference in change in systolic blood pressure level | Measured from baseline to 18 months
  The change in systolic blood pressure level from baseline to 18 months between the two arms.
Difference in change in diastolic blood pressure level | Measured from baseline to 18 months
  The change in diastolic blood pressure level from baseline to 18 months between the two arms.
Difference in change in total cholesterol level | Measured from baseline to 18 months
  The change in total cholesterol level from baseline to 18 months between the two arms.
Difference in change in low-density lipoprotein (LDL) cholesterol level | Measured from baseline to 18 months
  The difference in the change in LDL cholesterol level between the two arms.
Difference in change in fasting glucose level | Measured from baseline to 18 months
  The change in fasting glucose level from baseline to 18 months between the two arms.
Difference in change in hemoglobin A1c level | Measured from baseline to 18 months
  The change in hemoglobin A1c level from baseline to 18 months between the two arms
Difference in change in body weight | Measured from baseline to 18 months
  The change in body weight from baseline to 18 months between the two arms.
Appropriateness | Prior to baseline
  Percentage of participants, community health workers, providers, and church administrators who reply that the intervention is appropriate (good perceived fit). The outcome will be measured by survey question.
Adoption (provider) | At baseline
  Percentage of invited providers attending training sessions. Measured by study administrative data.
Adoption (church) | At baseline
  Percentage of churches adopting the intervention program. Measured by study administrative data.
Feasibility to participant, community health worker, provider and churches | Baseline
  Percentage of participants, community health worker, providers, and church administrators who reply that the intervention is feasible (actual fit, suitability). Measured by survey and study administrative data.
Acceptability | Measured at baseline, 6, 12, and 18 months
  Percentage of participants, community health worker, providers, and church administrators who reply that the intervention is acceptable (satisfactory). Measured by survey.
Penetrance (Participants) | Measured at baseline, 6, 12, and 18 months
  Percentage of enrolled participants receiving assigned intervention. Measured by study administrative data.
Costs | Baseline, 6, 12, and 18 months
  Implementation costs related to intervention and healthcare but not to study data collection. Measured by study administrative data.
Health Coaching Session Fidelity (community health worker-led strategy group) | Measured at 6, 12, and 18 months
  Percentage of health coaching sessions conducted. Measured by study administrative data.
Nutrition Education Session Fidelity (community health worker-led strategy group) | Measured at 6, 12, and 18 months
  Percentage of nutrition education sessions organized. Measured by study administrative data.
Exercise Session Fidelity (community health worker-led strategy group) | Measured at 6, 12, and 18 months
  Percentage of exercise sessions organized. Measured by study administrative data.
Health Care Appointment Fidelity (community health worker-led strategy group) | Measured at 6, 12, and 18 months
  Percentage of health care visit appointments made. Measured by study administrative data.
Penetrance (Providers) | Measured at baseline, 6, 12, and 18 months
  Percentage of trained providers delivering protocol-based care. Measured by study administrative data.
Penetrance (Educators) | Measured at baseline, 6, 12, and 18 months
  Percentage of trained CHWs or providers and health educators delivering health coaching. Measured by study administrative data.
Sustainability (Churches) | Measured at 24 months
  Percentage of churches continuing the intervention program and individual components. Measured by 6-month post-intervention survey.
Sustainability (Participants) | Measured at 24 months
  Percentage of participants maintaining ideal cardiovascular health metrics, healthy lifestyle components, and adherence to medications. Measured by 6-month post-intervention survey and examination.

OTHER OUTCOMES:
Difference in proportion of those receiving statin treatment who are eligible | Measured from baseline to 18 months
  Percentage of those receiving statin treatment who are eligible between the two arms over 18 months. Measured by survey data.
Difference in proportion of those who cease smoking of those who are current smokers at baseline | Measured from baseline to 18 months
  Percentage of those who cease smoking of those who are current smokers at baseline between the two arms over 18 months. Measured by survey data.
Difference in medication adherence | Measured from baseline to 18 months
  Percentage of self-reported medication adherence over 18 months. Self-reported medication adherence will be assessed using an medication adherence questionnaire.
Difference in quality of life (QoL) | Measured from baseline to 18 months
  The difference in QoL between the two arms over 18 months. QoL will be assessed using the SF-12 questionnaire. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Tulane University, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Our study data sharing plan will comply with all NIH policies for data sharing. Data sharing will be executed through the centralized NIH data repository and will be implemented in a timely manner. The study data, including data from baseline and follow-up visits, will be prepared for transmission to the NHLBI data repository - the Biologic Specimen and Data Repository Information Coordinating Center (BioLINCC). The datasets will be submitted to the NHLBI no later than three years after the end of the final participant follow-up or two years after the main paper of the trial has been published, whichever comes first. The NHLBI will review the submitted data prior to release. These data will be free of identifiers that allow identification of individual research participants either directly or through "deductive disclosure." In addition, we will offer, through our publicly accessible website, opportunities for outside investigators to collaborate with us using complete study data.
Supporting Information: Study Protocol, SAP
Time Frame: No later than three years after the end of the final participant follow-up or two years after the main paper of the trial has been published, whichever comes first

REFERENCES:
- [Background] Maroney K, Laurent J, Alvarado F, Gabor A, Bell C, Ferdinand K, He J, Mills KT. Systematic review and meta-analysis of church-based interventions to improve cardiovascular disease risk factors. Am J Med Sci. 2023 Sep;366(3):199-208. doi: 10.1016/j.amjms.2023.05.010. Epub 2023 May 25. PMID 37244637
- [Background] He J, Bundy JD, Geng S, Tian L, He H, Li X, Ferdinand KC, Anderson AH, Dorans KS, Vasan RS, Mills KT, Chen J. Social, Behavioral, and Metabolic Risk Factors and Racial Disparities in Cardiovascular Disease Mortality in U.S. Adults : An Observational Study. Ann Intern Med. 2023 Sep;176(9):1200-1208. doi: 10.7326/M23-0507. Epub 2023 Aug 15. PMID 37579311
- [Background] Bundy JD, Mills KT, He H, LaVeist TA, Ferdinand KC, Chen J, He J. Social determinants of health and premature death among adults in the USA from 1999 to 2018: a national cohort study. Lancet Public Health. 2023 Jun;8(6):e422-e431. doi: 10.1016/S2468-2667(23)00081-6. PMID 37244672